CLINICAL TRIAL: NCT05886998
Title: Nebulized Heparin for Prevention of Acute Lung Injury in Adult Patients Suffering Smoke Inhalation Injury: a Randomized Controlled Trial
Brief Title: Nebulized Heparin for Prevention of Acute Lung Injury in Smoke Inhalation Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh M. Hakim, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MD 238/2020
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-07

CONDITIONS: Smoke Inhalation Injury; Acute Lung Injury
Keywords: Smoke Inhalation Injury; Acute Lung Injury; Heparin
MeSH Terms: conditions — Smoke Inhalation Injury; Acute Lung Injury | interventions — Heparin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Nebulized Heparin) (Experimental): Heparin is nebulized via endotracheal tube
  Interventions: Drug: Heparin
- Group B (Nebulized Saline) (Placebo Comparator): Normal saline is nebulized via endotracheal tube
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Heparin — Heparin sodium (Generic, 5000 IU/ml ampoules)
  Arms: Group A (Nebulized Heparin)
Other: Normal Saline — 0.9% sodium chloride solution (normal saline)
  Other Names: Saline
  Arms: Group B (Nebulized Saline)

SUMMARY:
This study aims to examine the effects of nebulized heparin on the clinical outcomes in adult patients suffering smoke inhalation injury.

Patients will be randomized to receive nebulized heparin or an equal volume of normal saline for 14 days and the incidence of acute lung injury will be compared in either group.

DETAILED DESCRIPTION:
Adult patients who suffered smoke inhalation injury and who are candidates for elective intubation, have evidence of bronchial burn by fiberoptic bronchoscopy, have no evidence of acute lung injury and no more than 24 hours since inhalation injury will be included.

Patients will be randomized into 2 groups:

Group A (Intervention): Patients will receive 5000 IU heparin mixed with 3 ml saline and nebulized every 4 hours until they are extubated or until 14 days have elapsed whichever is earlier.

Group B (Control): Patients will receive 4 ml of normal saline nebulized every 4 hours until they are extubated or until 14 days have elapsed whichever is earlier.

The primary end point is the VFDs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients indicated for elective intubation:

* History of being trapped in a house or industrial fire.
* Production of carbonaceous sputum.
* Perioral facial burns affecting nose, lips, mouth, or throat .
* Altered level of consciousness at any time after the incident and including confusion.
* Symptoms of respiratory distress including a sense of suffocation, choking, breathlessness, and wheezing or discomfort affecting the eyes or throat, including irritation of the mucosal membranes.
* Signs of respiratory distress including stertorous or labored breathing, and tachypnea or auscultatory abnormalities, including crepitations or rhonchi.
* Hoarseness or loss of voice. 2. Evidence of bronchial burn by bronchoscopy to assess severity of inhalational trauma
* NO injury: absence of carbonaceous deposits, erythema, oedema, brochorrhea, or obstruction.
* Mild injury: minor patchy areas of erythema or carbonaceous deposits in proximal or distal bronchi.
* Moderate injury: moderate degree of erythema, carbonaceous deposits, bronchorrhea, or bronchial obstructions.
* Sever injury: sever inflammation with friability, copious carbonaceous deposits, bronchorrhea, or obstruction.
* Massive injury: evidence of mucosal sloughing, necrosis or endoluminal obliteration.

  3. No evidence of acute lung injury at presentation (either by radiology or ABG)
* Radiological findings: Normal lung without increased interstitial markings, ground glass opacification, or consolidation.
* ABG findings : PaO2/ Fio2 > 300. 4. Time between inhalational injury and intubation not longer than 24 hours.

Exclusion Criteria:

1. Burn injury > 24 hours.
2. History of pulmonary diseases.
3. Pregnancy or breast feeding.
4. History of allergy to heparin or HIT.
5. History or laboratory evidence of coagulopathy.
6. Burns area > 50% of total body surface area. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
VFDs | 28 days
  Number of days free of mechanical ventilation

SECONDARY OUTCOMES:
ICU-free days | 28 days
  Number of days free from ICU and alive
Duration of mechanical ventilation | 28 days
  Time from institution to termination of mechanical ventilation
Mortality | 28 days
  Survival to ICU discharge
Side effects | 28 days
  Occurrence of heparin-induced adverse effects, e.g., thrombocytopenia, abnormal bleeding
P/F ratio | 14 days
  PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M Hakim, MD, Principal Investigator — Ain Shams University Faculty of Medicine
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424